CLINICAL TRIAL: NCT03317730
Title: Pilot Trial of Microsphere Oxycodone (Xtampza ER) for Pain Management in Patients Receiving Radiotherapy for Locally Advanced Head and Neck Cancer
Acronym: RAD 1702
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Andrew McDonald, Assistant Professor - Department of Radiation Oncology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300000574
Record Dates: First submitted 2017-10-11; First posted 2017-10-23 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Locally Advanced Head and Neck Cancer
Keywords: Xtampza ER; LAHNC; Head and neck cancer; Pain management
MeSH Terms: conditions — Head and Neck Neoplasms; Agnosia | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RT + Xtampza ER (Experimental): This study will enroll patients scheduled to receive radiation therapy (RT), but RT details are not specified by this protocol. Patients taking long acting opioid analgesics prior to enrollment will be converted to an equivalent dose of Xtampza ER at the time of enrollment. For the remaining patients not previously prescribed opioid analgesics, Xtampza ER will be initiated when 2 or more daily doses of short acting opioids are required, resulting in a total daily dose of at least 30mg morphine sulfate equivalent. During RT, pain will be assessed on a weekly basis using the PI-NRS and the dose of Xtampza ER will be adjusted at the discretion of the treating physician, with recommendation to maintain an equivalent of 100% daily opioid requirement. Assessment for tapering of Xtampza ER will begin 1 month following the completion of RT at the time of first follow-up.The study period will end 3 months following the final fraction of RT.
  Interventions: Drug: Xtampza ER

INTERVENTIONS:
Drug: Xtampza ER — Xtampza ER is a wax microsphere formulation of oxycodone that results in a nearly identical pharmacokinetic profile regardless of whether the capsule is intact when ingested or if ingested via enteral feeding tube as opposed to by mouth.

SUMMARY:
To confirm the feasibility of studying Xtampza ER during radiotherapy (RT) for LAHNC as part of a prospective clinical trial.

DETAILED DESCRIPTION:
To confirm the feasibility of studying Xtampza ER during radiotherapy (RT) for locally advanced head and neck cancer (LAHNC) as part of a prospective clinical trial. Investigators will also assess pain control, quality of life, and drug related toxicity during RT and during short term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced cancer of mucosa of the head and neck.
* Eligible subsites will include nasal cavity, paranasal sinuses, nasopharynx, oropharynx, oral cavity, major salivary glands, oropharynx, larynx, hypopharynx, cervical esophagus, or unknown primary site with lymph node metastases.
* Clinical or pathologic stage III-IV
* Scheduled to receive RT with curative intent with the expectation that some portion of the mucosa of the upper aerodigestive tract will receive a dose of at least 50 Gray.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Age > 19 years
* Subjects given written informed consent

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Feasibility of Xtampza ER during radiotherapy (RT) for locally advanced head and neck cancer (LAHNC). | 1 year
  Feasibility of administering Xtampza ER during RT is defined as continuation of the medication throughout RT. The number of patients who discontinue Xtampza ER due to difficulty with administration, perceived inefficacy, or toxicity will be recorded.

SECONDARY OUTCOMES:
Determine Pain Control (at time of enrollment) | 1 year
  Pain will be assessed using:
  Pain Intensity Numeric Rating Scale - a scale of 0-10, with 0 being no pain and 10 being worst possible pain.
  Brief Pain Inventory - a patient completed 2-page questionnaire rating severity of pain and how pain interferes with functioning. The pain severity score is calculated by averaging the 4 questions related to this topic (each question is a 0-10 scale, with higher numbers indicating worse pain). The pain interference score is calculated by averaging the 7 questions related to this topic (each question is a 0-10 scale, with higher numbers indicating worse functional interference). The remaining items included in the Brief Pain Inventory will be recorded but do not contribute to a score.
Determine Pain Control (weekly during RT) | 1 year
  Pain will be assessed using:
  Pain Intensity Numeric Rating Scale - a scale of 0-10, with 0 being no pain and 10 being worst possible pain.
  Brief Pain Inventory - a patient completed 2-page questionnaire rating severity of pain and how pain interferes with functioning. The pain severity score is calculated by averaging the 4 questions related to this topic (each question is a 0-10 scale, with higher numbers indicating worse pain). The pain interference score is calculated by averaging the 7 questions related to this topic (each question is a 0-10 scale, with higher numbers indicating worse functional interference). The remaining items included in the Brief Pain Inventory will be recorded but do not contribute to a score.
Determine Pain Control (at follow-up) | 1 year
  Pain will be assessed using:
  Pain Intensity Numeric Rating Scale - a scale of 0-10, with 0 being no pain and 10 being worst possible pain.
  Brief Pain Inventory - a patient completed 2-page questionnaire rating severity of pain and how pain interferes with functioning. The pain severity score is calculated by averaging the 4 questions related to this topic (each question is a 0-10 scale, with higher numbers indicating worse pain). The pain interference score is calculated by averaging the 7 questions related to this topic (each question is a 0-10 scale, with higher numbers indicating worse functional interference). The remaining items included in the Brief Pain Inventory will be recorded but do not contribute to a score.
Access Toxicity | 1 year
  Toxicity will be assessed using the Common Terminology Criteria for Adverse Events version 4.03. Assessments will be at time of enrollment, weekly during RT, and at follow-up.
Access Quality of Life | 1 year
  The FACT - Head & Neck questionnaire will be administered at time of enrollment, completion of RT, and at follow-up.
  The FACT - Head & Neck questionnaire is a battery of 39 questions across 5 domains, with each response given on a 0-4 scale, with 0 indicating no problem and 4 indicating severe problem. The average of responses within each domain will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Hazelrig-Salter Radiation Oncology Center, Birmingham, Alabama, United States